CLINICAL TRIAL: NCT03344367
Title: A Phase 1, Open-Label Study of JWCAR029, CD19-targeted Chimeric Antigen Receptor (CAR) T Cells, for Adult Subjects With Relapsed and Refractory (R/R) B-cell Non-Hodgkin Lymphoma (NHL)
Brief Title: Study Evaluating the Safety and Efficacy of JWCAR029 in Adult Subjects With Relapsed and Refractory B-cell Non-Hodgkin Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Collaborators: Shanghai Mingju Biotechnology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Jun Zhu, Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR029-001
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Non Hodgkin Lymphoma
Keywords: Non Hodgkin Lymphoma; CD19-targeted chimeric antigen receptor; JWCAR029
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — relmacabtagene autoleucel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JWCAR029 (Experimental): The safety and efficacy of JWCAR029 will be evaluated in a standard 3+3 dose escalation approach. 5 CAR T dosage will be tested in this study: 1×10^7, 2.5×10^7, 5×10^7, 1×10^8, 1.5^108 CAR+ T cells.
  Interventions: Biological: JWCAR029

INTERVENTIONS:
Biological: JWCAR029 — Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of JWCAR029. During JWCAR029 production, subjects will receive a conditioning chemotherapy regimen of cyclophosphamide and fludarabine for the purpose of lymphocytes depletion. After lymphodepletion, subjects will receive one dose treatment with JWCAR029 by intravenous (IV) injection.

SUMMARY:
This is a single arm, open-label, dose escalation clinical study to evaluate the safety and efficacy of infusion of autologous CD19-targeted chimeric antigen receptor (CD19 CAR) T cells in adult subjects with relapsed and refractory B-cell Non-Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be enrolled in this study:

  1. Age ≥ 18 years at the time of consent
  2. Signed written informed consent obtained prior to any study procedures
  3. Relapsed or refractory B-cell NHL.
  4. PET-positive disease BY Lugano classification
  5. Archived tumor biopsy tissue available from the last relapse and corresponding pathology report available or, if at least one tumor-involved site is deemed accessible at time of screening, willing to undergo pre-treatment biopsy (excisional when possible) for disease confirmation. If a subject has never had a complete response, a sample from the most recent biopsy is acceptable.
  6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
  7. Adequate bone marrow, renal, hepatic, pulmonary and cardiac function
  8. Adequate vascular access for leukapheresis procedure
  9. Subjects who have received previous CD19-targeted therapy must have CD19-positive lymphoma confirmed on a biopsy since completing the prior CD19-targeted therapy
  10. Subjects must agree to use appropriate contraception.

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from participation in this study:

  1. Subjects with central nervous system (CNS)-only involvement by malignancy (note: subjects with secondary CNS involvement are allowed on study)
  2. History of another primary malignancy that has not been in remission for at least 2 years.
  3. Treatment with alemtuzumab within 6 months of leukapheresis, or treatment with fludarabine or cladribine within 3 months of leukapheresis
  4. Active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection at the time of screening
  5. Subjects with uncontrolled systemic fungal, bacterial, viral or other infection despite appropriate antibiotics or other treatment at the time of leukapheresis or JWCAR029 administration
  6. Presence of acute or chronic graft-versus-host disease (GVHD)
  7. History of cardiovascular disease
  8. History or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
  9. Pregnant or nursing women.
  10. Prior CAR T-cell or other genetically-modified T-cell therapy, with the exception of prior JWCAR029 treatment in this protocol for subjects receiving retreatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-16 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse events (AEs) | 2 years
  Physiological parameter
Dose-limiting toxicities of JWCAR029 | 28 days after JWCAR029 infusion
  Physiological parameter
Objective response rate (ORR) | 2 years
  Lugano criteria

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of JWCAR029 in the peripheral blood and bone marrow | 1 year after JWCAR029 infusion
  Flow cytometry and qPCR
Time to maximum concentration (Tmax) of JWCAR029 in the peripheral blood and bone marrow | 1 year after JWCAR029 infusion
  Flow cytometry and qPCR
Area-under the concentration-vs-time-curve (AUC) of JWCAR029 in the peripheral blood and bone marrow | 1 year after JWCAR029 infusion
  Flow cytometry and qPCR
Complete response (CR) rate | 2 years
  Lugano criteria
Duration of response | 2 years
  Lugano criteria
Progression-free survival (PFS) and PFS ratio | 2 years
  Lugano criteria
Overall survival | 2 years
  Physiological parameter
Health-related quality of life (HRQoL) | 2 years
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338